CLINICAL TRIAL: NCT02601781
Title: A Prospective Evaluation of a Standardized Strategy for the Use of Bioresorbable Vascular Scaffold in ST-segment Elevation Myocardial Infarction: the BVS STEMI STRATEGY-IT Registry
Brief Title: Use of BVS in ST-segment Elevation Myocardial Infarction (STEMI): the BVS STEMI STRATEGY-IT Prospective Registry
Acronym: STRATEGY-IT
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Azienda Ospedaliera Bolognini di Seriate Bergamo (Other)
Responsible Party: Principal Investigator, Alfonso Ielasi, MD, Azienda Ospedaliera Bolognini di Seriate Bergamo
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AOBolognini
Record Dates: First submitted 2015-10-16; First posted 2015-11-10 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: ST-elevation Myocardial Infarction (STEMI)
Keywords: Bioresorbable Vascular Scaffold (BVS); STEMI; Primary PCI
MeSH Terms: conditions — ST Elevation Myocardial Infarction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Primary PCI (PPCI) with BVS (Experimental): Primary percutaneous coronary intervention (PPCI) with bioresorbable vascular scaffold (BVS) implantation in STEMI patients. Following the arterial route, PPCI (performed according to the international guidelines) aims to recanalize an occluded coronary artery that is then maintained patent inserting an endovascular permanent prosthesis (stent). In this study we aim to assess the results following the use of a fully bioresorbable prosthesis (BVS) during PPCI using a pre-specified implantation strategy (eventual thrombectomy, intravascular imaging, lesion pre-dilatation, BVS implantation and BVS post-dilatation). BVS has the theoretical advantage, as compared with a permanent stent, to disappear within 24-36 months from implantation restoring the native pristine vessel state.
  Interventions: Procedure: Primary percutaneous coronary intervention (PPCI); Device: Bioresorbable Vascular Scaffold (BVS ABSORB)

INTERVENTIONS:
Procedure: Primary percutaneous coronary intervention (PPCI) — Primary percutaneous coronary intervention (PPCI) aims to recanalize an occluded coronary artery causing ST-elevation myocardial infarction (STEMI).
Device: Bioresorbable Vascular Scaffold (BVS ABSORB) — BVS Use during Primary PCI following a pre-specified implantation strategy (eventual thrombectomy, intravascular imaging, lesion pre-dilatation, BVS implantation and BVS post-dilatation).

SUMMARY:
BVS STEMI STRATEGY-IT is a spontaneous, prospective, non-randomized, single-arm multicenter registry on consecutive STEMI patients eligible to undergo primary percutaneous coronary intervention (PPCI) with BVS implantation on the basis of the pre-specified inclusion and exclusion criteria.

This registry has the objective to assess the immediate (peri-procedural and 30 days), mid (6 months and 1 year) and long-term (3 and 5 years) results following BVS implantation using a pre-specified implantation strategy during PPCI in STEMI subjects.

DETAILED DESCRIPTION:
Population:

This registry is intended to obtain data from consecutive STEMI patients undergoing PPCI with BVS implantation in 10-15 Italian sites.

STEMI is defined according to the European guidelines criteria.

Procedure:

Dual Anti-Platelet and Antithrombotic Regimen:

Patients undergoing PPCI should receive a combination of aspirin (i.v. or os) and a loading dose of oral P2Y12 receptor blocker (ticagrelor, prasugrel or clopidogrel only when prasugrel or ticagrelor are not available or are contraindicated) as early as possible before angiography and a parenteral anticoagulant according to the current guidelines. In particular the early administration (at least just outside the cath-lab or at first medical contact/ambulance in case of ticagrelor) of the P2Y12 receptor blocker loading dose (ticagrelor 180 mg, prasugrel 60 mg or clopidogrel 600 mg when prasugrel or ticagrelor are not available or are contraindicated) could be of paramount importance when a BVS is implanted in a thrombotic setting to reduce the risk of device thrombosis. For this reason, in case of angiographic evidence of large thrombus the use of a glycoprotein should be considered according to the current guidelines.

The P2Y12 inhibitor recommended (ticagrelor 90 mg bid, prasugrel 10 mg or clopidogrel 75 mg) in addition to acetyl salicylic acid should be maintained for at least 12 months after BVS implantation (with the decision for longer term use left to the discretion of the treating physician according to the specific clinical scenario). Anticoagulation is recommended for all patients in addition to anti-platelet therapy during PPCI according to the current guidelines.

Access Site:

Even if no specific arterial site access is mandatory, the radial approach should be the preferred method of access.

Guiding Catheter and Guide-wires:

The guiding catheter and the guide-wires should be choose (both according to each Institution preference) to obtain the maximum stability of the system and to facilitate the BVS delivery to the culprit site. The use of 6 Fr guiding catheters is recommended even if BVS (2.5 and 3.0) can also be implanted via 5 Fr guiding catheters.

BVS Size Selection BVS sizes actually available are limited (diameter: 2.5 mm, 3.0 mm, 3.5 mm and length: 8, 12 mm, 18 mm, 23 mm and 28 mm). In order to reduce the vasoconstriction typical of the STEMI setting and to accurately select the BVS diameter is fundamental to obtain the maximum vessel dilatation by the administration of intracoronary bolus of vasodilator drugs (i.e. nitroglycerin or adenosine) after TIMI flow (>0) restoration. Once maximal dilatation is obtained (vasodilators drugs strongly recommended), the BVS size selection should be made accordingly to the maximal vessel diameter (visually estimated by the operator) assessed immediately proximal and distal to the culprit lesion site (in 2 orthogonal angiographic views). This step is of paramount importance considering the maximal post-expansion BVS limit (+0.5 mm vs. the nominal BVS diameter) as compared to the newer generation DES (1.0 mm vs. the nominal DES diameter). For this reason a slight BVS diameter overestimation compared to the visually estimated reference vessel size is suggested (i.e. BVS 3.5 mm for a reference vessel diameter [RVD]> 3.0 mm, BVS 3.0 mm for a RVD>2.5 mm).

As compared to visual estimation, quantitative coronary angiography (QCA) provides more objective information even if it also tends to underestimate the lumen diameter. Intracoronary imaging systems such as intravascular ultrasound (IVUS) or optical coherence tomography (OCT) may help to overcome the aforementioned limitations and may be considered an important tool for scaffold size selection. Even if intravascular imaging use is not routinely required in this study it can be performed at operator's discretion.

Pre-dilatation:

Lesion preparation before deployment is an essential step for patients receiving BVS, where the goal of lesion preparation is to facilitate scaffold delivery, reduce plaque shift, and, most importantly, to allow optimal scaffold expansion.

BVS Implantation:

Prior to use, the everolimus-eluting BVS system will be inspected and prepared according to the Instruction for Use (IFU). The BVS should cover 2-5 mm of the healthy vessel at either edge of the culprit lesion. BVS deployment must be performed gradually, inflating the delivery system's balloon in 2 atm increments (up to the rated burst pressure) every five seconds until complete expansion of the BVS. Once reached, the target pressure is maintained (if tolerated by the patient) for at least 30 seconds to favour the device expansion. Multiple BVS overlapping is allowed in case of long lesion involving the culprit site. However the thick BVS struts mandate to minimize the overlapping length particularly in the STEMI setting. If overlap is required starting with the distal scaffold is preferred except in case a proximal landmark (i.e. long lesion involving the ostial segment of the vessel) must be respected. Among the different BVS overlapping strategies proposed19, the marker-to-marker (the second more proximal BVS is advanced until the distal balloon markers line up with the proximal marker beads of the implanted scaffold obtaining about 1 mm of struts overlap) technique is that suggested in this study. Use of angiographic "stent enhancement" tool in two orthogonal projections can help the marker-to-market positioning. A "hybrid" BVS-DES overlapping is not allowed. In case of culprit lesions involving a bifurcation site, a single-BVS approach (after wire positioning in the side branch ["keep it open"]) and nothing else is suggested. In case of flow-limiting thrombus shift from the main to the side-branch (SB), consider a BVS fenestration toward the SB with a semi-compliant balloon (2.0-3.0 mm diameter according to the SB dimension). If a second device is required as a bail-out strategy (i.e. persistent flow limitation after balloon dilatation at the SB), a metallic stent implantation should be considered. In case of bifurcated culprit lesions where a 2-stent strategy is planned as intention-to-treat it is advisable to avoid BVS implantation.

In case of extensive CAD in vessels remote (multi-vessel CAD) from the infarct-related artery, the culprit lesion only should be systematically treated during the initial intervention. Immediate (preventive) intervention in non-infarct-related lesions is not recommended. In this case, staged PCI should be performed within 50 days after PPCI while BVS implantation is suggested in order to complete the revascularization according to the lesion characteristics.

Post-dilatation:

BVS deployment in the STEMI setting should aim to: 1) obtain full BVS expansion with less than 20% residual stenosis at the culprit site; 2) reduce distal embolization (slow-flow/no-reflow phenomenon) taking advantage of the BVS strut thickness (so called "snow-racket concept"). Even if post-dilatation is not routinely performed during PPCI with new generation intracoronary prosthesis (15-20% of the cases), it may be required (and encouraged in this study) after BVS implantation in STEMI patients. In particular the inflation of a non-compliant balloon (for 10-60 seconds if tolerated by the patient) with a maximum diameter 0.5 mm more than the BVS diameter is suggested in case of TIMI 3 flow and more than 20% residual stenosis (by angiographic visual estimation). In case of TIMI 3 flow and less than 20% residual stenosis the decision to post-dilate (with a NC balloon with the same nominal diameter of BVS implanted) is left at operator's discretion. Post-dilatation could be avoided in case of: 1) no residual stenosis associated with adequate BVS expansion and apposition (preferably confirmed by intravascular imaging systems -IVUS or OCT-); 2) transient slow-flow or no-reflow during BVS implantation with subsequent TIMI flow 3 restoration.

Follow-up:

Clinical data will be collected by the medical staff of each participating center by hospital visit or telephone contact at 30 days, 6 months, 1 year, 3-and 5-years after PPCI. Angiographic follow-up is not mandatory but performed only in case of planned "step" revascularisation or if clinically indicated at follow-up. However, patients undergoing angiographic follow-up (and IVUS or OCT follow-up) will be included in subgroup analysis.

Data Collection:

Clinical, lesion, procedural data and follow-up outcomes of patients who have given a written informed consent are entered into a web-based Case Report Form (CRF). The monitoring of the study and the data entry will be continuously supervised by the Steering Committee in order to respect the enrollment plan.

Enrolment:

The enrolment period is limited to 12 months since the first patient is enrolled in the specific participating center. However it could be extended if recruiting proceeds slowly.

Informed Consent and Withdrawal criteria:

All the patients must sign a written informed consent to be enrolled in the registry.

The patient has the right to withdraw from the registry at any time and without reason. Upon early withdrawal from the registry, the case report form (CRF) should be completed as far as possible and the reasons for withdrawal should if possible be documented.

Statistical Methods:

Numerical data will be presented as the mean ± standard deviation and minimum and maximum values. Categorical data will be presented as counts and percentages of the total. Cross tabulations and subgroup summary statistics will be calculated where necessary. Two-sided 95% confidence intervals will be given where adequate. All data are presented using descriptive statistical methods. For metric data sets, the mean values, standard deviation, median, maximum and minimum as well as the 95% confidence interval are stated. For categorical data, absolute and relative frequencies are determined, and the exact 95% confidence interval is calculated. Furthermore, for primary and secondary end-points, Kaplan Meier curves will be presented and event-free survival analysis will be performed to compare subgroups.

Sample Size Justification:

The paper of Brugaletta et al. (BVS-EXAMINATION) reported an incidence of DOCE of 3.1% at 30 days: given the potential important impact of a pre-specified implantation strategy in STEMI patients undergoing BVS implantation, and aiming to appraise a reduction to 0.7%, 505 patients are required to have a 80% chance of detecting, as significant at the 5% level, a decrease in the primary outcome of 2.4%. (Pocock SJ. Clinical Trials: A Practical Approach. Wiley; 1983) The paper of Brugaletta et al. (BVS-EXAMINATION) reported an incidence of DOCE of 3.1% at 30 days (9/290). Accordingly, the Investigators computed that a target sample of 500 patients will enable the computation of reasonably precise 95% confidence intervals. Specifically, assuming the rate of 3.1% DOCE at 30 days, confidence intervals computed with the Welson score would be from 2% to 5.1% (16/500).

Confidentiality:

The investigator shall maintain patient confidentiality during all audits and inspections of the clinical site and documentation. Registry patients will be identified only by a unique patient number, used in correspondence and on the registry database. The Investigator will keep a list in which each patient is named along with their assigned patient number.

ELIGIBILITY:
Inclusion Criteria:

1. Patients presenting with a ST-elevation myocardial infarction (STEMI) with symptoms onset <12 hours from hospital admission eligible for PPCI and BVS implantation;
2. Signed Patient Informed Consent/Data Release Form.

Exclusion Criteria:

1. Age >75 years or <18 years;
2. Cardiogenic shock;
3. Pregnancy or breastfeeding;
4. Infarct-artery max diameter (within planned device deployment segment) <2.5 or >3.7 mm;
5. Stent thrombosis/restenosis as a culprit lesion;
6. Acute occlusion of a saphenous vein graft as a culprit lesion;
7. Culprit lesion involving a bifurcation which requires a 2-stent strategy as intention-to-treat;
8. Culprit lesion involving a long diseased segment requiring hybrid (overlap BVS-DES) treatment;
9. Dialysis;
10. Comorbidities with life expectancy <3 years;
11. Contraindication to 12 months dual anti-platelet therapy;
12. Severe calcification or/tortuosity in the segments proximal to the culprit lesion;
13. Absolute indication to chronic anticoagulation therapy;
14. Elective or emergent cardiac surgery intervention within 1 year after PPCI (i.e. inferior STEMI with critical unprotected left main disease or mechanical complications of STEMI).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Actual)
Dates: Start 2015-10; Primary Completion 2016-12 (Actual); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Device oriented composite end-point (DOCE) | 30 days
  A device oriented composite end-point of cardiac death, any myocardial infarction (STEMI or NSTEMI) clearly attributable to the-intervention culprit vessel (TV-MI) and ischemic driven TLR within 30 days after the index procedure.

SECONDARY OUTCOMES:
Procedural Success | 0-7 days
  Procedural success defined as BVS implantation at the "culprit" lesion site with less than 20% final stenosis and distal TIMI 3 flow.
Device oriented composite end-point (DOCE) | 6 months; 1, 3, 5 years
  A device oriented composite end-point (cardiac death, any myocardial infarction [STEMI or NSTEMI] clearly attributable to the-intervention culprit vessel [TV-MI] and ischemic driven TLR) at 6 months, 1-, 3-, and 5-years follow-up.
BVS Thrombosis | In Hospital and at follow-up (up to 5 years)
  Any Definite/Probable BVS thrombosis (in-hospital and at follow-up).
Any Bleeding | In Hospital and at follow-up (up to 5 years)
  Bleedings defined according to the Bleeding Academic Research Consortium (BARC)
Major adverse cardiovascular events (MACE) | In Hospital and at follow-up (up to 5 years)
  Cardiac death, any TV-MI, target vessel revascularization (TVR) and TLR in-hospital or at follow-up;
ST-segment resolution at the electrocardiogram (ECG) | 60 minutes
  ST-segment resolution at ECG within 60 minutes of primary PCI.

CONTACTS AND LOCATIONS:
Overall Officials: Alfonso Ielasi, MD, Principal Investigator — Azienda Ospedaliera Bolognini di Seriate Bergamo
Locations (1):
- Cardiology Division, Azienda Ospedaliera Bolognini Seriate, Seriate (BG), Italy

REFERENCES:
- [Background] Ielasi A, Varricchio A, Campo G, Leoncini M, Cortese B, Vicinelli P, Brugaletta S, di Uccio FS, Latib A, Tespili M. A prospective evaluation of a standardized strategy for the use of a polymeric everolimus-eluting bioresorbable scaffold in ST-segment elevation myocardial infarction: Rationale and design of the BVS STEMI STRATEGY-IT study. Catheter Cardiovasc Interv. 2017 Jun 1;89(7):1129-1138. doi: 10.1002/ccd.26801. Epub 2016 Oct 24. PMID 27774758
- [Result] Cortese B, Ielasi A, Romagnoli E, Varricchio A, Cuculo A, Loi B, Pisano F, Corrado D, Sesana M, La Vecchia L, Summaria F, Tespili M, Silva Orrego P, Tognoni G, Steffenino G. Clinical Comparison With Short-Term Follow-Up of Bioresorbable Vascular Scaffold Versus Everolimus-Eluting Stent in Primary Percutaneous Coronary Interventions. Am J Cardiol. 2015 Sep 1;116(5):705-10. doi: 10.1016/j.amjcard.2015.05.049. Epub 2015 Jun 3. PMID 26100584
- [Result] Ielasi A, Cortese B, Varricchio A, Tespili M, Sesana M, Pisano F, Loi B, Granata F, Moscarella E, Silva Orrego P, La Vecchia L, Steffenino G; RAI registry investigators. Immediate and midterm outcomes following primary PCI with bioresorbable vascular scaffold implantation in patients with ST-segment myocardial infarction: insights from the multicentre "Registro ABSORB Italiano" (RAI registry). EuroIntervention. 2015 Jun;11(2):157-62. doi: 10.4244/EIJY14M10_11. PMID 25354760
- [Result] Brugaletta S, Gori T, Low AF, Tousek P, Pinar E, Gomez-Lara J, Scalone G, Schulz E, Chan MY, Kocka V, Hurtado J, Gomez-Hospital JA, Munzel T, Lee CH, Cequier A, Valdes M, Widimsky P, Serruys PW, Sabate M. Absorb bioresorbable vascular scaffold versus everolimus-eluting metallic stent in ST-segment elevation myocardial infarction: 1-year results of a propensity score matching comparison: the BVS-EXAMINATION Study (bioresorbable vascular scaffold-a clinical evaluation of everolimus eluting coronary stents in the treatment of patients with ST-segment elevation myocardial infarction). JACC Cardiovasc Interv. 2015 Jan;8(1 Pt B):189-197. doi: 10.1016/j.jcin.2014.10.005. PMID 25616924
- [Derived] Ielasi A, Campo G, Cortese B, Leoncini M, Varricchio A, Brugaletta S, Favaretto E, Fineschi M, Piraino D, Calabria P, Granata F, Pisano F, Mussardo M, Latib A, Tespili M. One-Year Results Following a Pre-Specified ABSORB Implantation Strategy in ST-Elevation Myocardial Infarction (BVS STEMI STRATEGY-IT Study). Cardiovasc Revasc Med. 2019 Aug;20(8):700-704. doi: 10.1016/j.carrev.2018.10.003. Epub 2018 Oct 4. PMID 30314835
- [Derived] Ielasi A, Campo G, Rapetto C, Varricchio A, Cortese B, Brugaletta S, Geraci S, Vicinelli P, Scotto di Uccio F, Secco GG, Poli A, Nicolini E, Ishida K, Latib A, Tespili M. A Prospective Evaluation of a Pre-Specified Absorb BVS Implantation Strategy in ST-Segment Elevation Myocardial Infarction: The BVS STEMI STRATEGY-IT Study. JACC Cardiovasc Interv. 2017 Sep 25;10(18):1855-1864. doi: 10.1016/j.jcin.2017.07.023. PMID 28935077